CLINICAL TRIAL: NCT03801382
Title: Study to Establish the Psychometric Properties of the Digital Cognitive Tests on the Philips IntelliSpace Cognition Platform
Brief Title: Psychometric Properties of IntelliSpace Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Collaborators: Research America Inc. (Industry); Qserve (Industry); Factory CRO (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ICBE-2-28674
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Functioning of Healthy Individuals
Keywords: cognitive model; cognitive assessment; digital cognitive tests; automated scoring; algorithms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (5):
- Digital / Paper (Other): Phase 1: Participants' cognition is measured using digital tests. Phase 2: Participants' cognition is measured using paper-pencil tests.
  Interventions: Device: IntelliSpace Cognition (ISC); Diagnostic Test: Paper-Pencil Tests
- Paper / Digital (Other): Phase 1: Participants' cognition is measured using paper-pencil tests. Phase 2: Participants' cognition is measured using digital tests.
  Interventions: Device: IntelliSpace Cognition (ISC); Diagnostic Test: Paper-Pencil Tests
- Digital / Digital (Other): Phase 1: Participants' cognition is measured using digital tests. Phase 2: Participants' cognition is measured using digital tests.
  Interventions: Device: IntelliSpace Cognition (ISC)
- Paper / Paper (Other): Phase 1: Participants' cognition is measured using paper-pencil tests. Phase 2: Participants' cognition is measured using paper-pencil tests.
  Interventions: Diagnostic Test: Paper-Pencil Tests
- Digital (Other): Phase 1: Participants' cognition is measured using digital tests. Phase 2: N/A
  Interventions: Device: IntelliSpace Cognition (ISC)

INTERVENTIONS:
Device: IntelliSpace Cognition (ISC) — Philips ISC is a Class-II Medical Device in the US and provides objective data regarding cognition via scoring algorithms that HCPs can use to inform diagnostic decision making and treatment planning. It enables tracking cognition over time and offers the possibility of new outcome measures. ISC can be used in a variety of healthcare environments such as neurology and neuropsychology practices.
  Arms: Digital; Digital / Digital; Digital / Paper; Paper / Digital
Diagnostic Test: Paper-Pencil Tests — The same cognitive tests that are on the ISC platform are performed using paper and pencil (rather than digitally) as is the case in standard clinical practice.
  Arms: Digital / Paper; Paper / Digital; Paper / Paper

SUMMARY:
This study aims to validate the tests that are on the IntelliSpace Cognition platform and to establish normative data for these tests.

ELIGIBILITY:
Inclusion Criteria:

* Examinee's primary language (language most often spoken) must be English.
* If examinee has vision impairment or hearing loss, must be corrected to normal.
* Must have normal fine and gross motor ability
* Must have use of fingers, hands, and arms to be able to use a pencil to write symbols.
* Must be able to understand subtest instructions and participate fully in testing.

Exclusion Criteria:

* Evidence of current cognitive impairment.
* Disruptive behavior or insufficient compliance with testing to ensure a valid assessment.
* Examinee must not be currently admitted to a hospital, assisted living, nursing home or a psychiatric facility.
* Examinee must not be diagnosed with a neurological disorder or disease (e.g., Parkinson's, brain tumor, stroke, TBI, epilepsy [if # seizures ≤ 2 and not receiving ongoing treatment for seizures, and not currently seeking medical evaluation or attention related to seizures, examinee can be accepted], encephalitis, dementia, language disorder (expressive or mixed receptive/expressive excluded; articulation disorder is ok), learning disorder.
* Must not have been unconscious related to traumatic brain injury or "medical condition" > 20 minutes (however, e.g., heat stroke, medication induced are ok) or any head-injury resulting in an overnight hospital stay.
* Any history of a medical event requiring resuscitation in which examinee was non-responsive for > 15 minutes.
* Must not have current or recent functional change (ability to carry out usual duties at work, in school, IADLs [driving, shopping, managing money], etc.) due to cognitive change.
* Examinee must not be receiving chemotherapy treatment, or have received chemotherapy treatment in the past 2 months.
* Examinee must not have a history of ECT or radiation to the CNS.
* Examinee must not be (currently or in the past) diagnosed with a psychotic disorder, or currently diagnosed with a mood disorder (however, Major Depressive Disorder in remission or with no current episode, and Dysthymic and Adjustment Disorders, are acceptable) or an anxiety disorder with symptoms significant enough to interfere with optimal test performance.
* Autoimmune disorder (e.g., LUPUS, Multiple Sclerosis)
* Examinee must not be currently diagnosed with substance abuse or dependence, or have carried any substance abuse or dependence diagnosis in the past year (> 1 year in remission diagnoses are ok). Long term alcohol abusers are excluded as well (e.g., abused substance for more than 10 years).
* Any history of Autism Spectrum Disorder or Intellectual Disability.
* The examinee must not be currently taking medication that might impact test performance (e.g., anti-convulsants, antipsychotics, benzodiazepines, psychostimulants, opiods, tricyclic antidepressants, some norepinephrine reuptake inhibitors). Most antihypertensive medications and statins are acceptable.
* If previously diagnosed with any physical condition or illness that might depress test performance, illness must not interfere with normal cognitive functioning at work, school, ADLs, etc. Diabetes, hypothyroidism, and hypertension are acceptable if controlled.
* Exclude primarily nonverbal or uncommunicative. Must not have a diagnosis of aphasia.
* Examinees should not have received neuropsychological testing although previous MMSE testing is allowed if more than 6 months prior
* Examinee must not be seeking medical diagnostic procedures for cognitive difficulties from a medical professional.
* Non-valid health insurance in USA.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research America Inc., Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: First Assessment
Arm/Group | Digital / Paper | Paper / Digital | Digital / Digital | Paper / Paper | Digital
Started | 99 | 101 | 53 | 49 | 148
Completed | 99 | 101 | 53 | 49 | 148
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Second Assessment
Arm/Group | Digital / Paper | Paper / Digital | Digital / Digital | Paper / Paper | Digital
Started | 99 | 101 | 53 | 49 | 0
Completed | 99 | 101 | 53 | 49 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Digital / Paper | Paper / Digital | Digital / Digital | Paper / Paper | Digital | Total
Number analyzed (Participants) | 99 | 101 | 53 | 49 | 148 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (7) | 66.3 (7.5) | 65.9 (7.4) | 65.7 (7.3) | 62 (8.9) | 64.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 53 | 29 | 27 | 79 | 238
  Male | 49 | 48 | 24 | 22 | 69 | 212
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 5 | 6 | 14 | 40
  Not Hispanic or Latino | 93 | 92 | 48 | 43 | 134 | 410
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 99 | 101 | 53 | 49 | 148 | 450
MMSE [Mean (Standard Deviation); unit: units on a scale] — Mini-Mental State Examination The MMSE has a scale that ranges from 0 to 30 with higher scores indicating a better outcome.
  units on a scale | 27.6 (1.9) | 27.6 (2.1) | 27.1 (1.9) | 27.9 (1.6) | 27.8 (1.7) | 27.6 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Scores Digital (ISC) Tests
Description: Scores retrieved from all cognitive tests on the ISC platform The cognitive tests included on the ISC platform are commonly used in neuropsychological assessments and measure aspects of executive functioning (TMT A, TMT B, Star Cancellation Test, RAVLT, Letter Fluency Test, Category Fluency Test, ROCFT, Digit Span Forward, Digit Span Backward), processing speed (Star Cancellation Test), working memory (TMT A, TMT B, Star Cancellation Test, Letter Fluency Test, Digit Span Forward, Digit Span Backward), memory (RAVLT), verbal processing (Letter Fluency Test, Category Fluency Test), and visual-spatial processing (RAVLT, ROCFT).
Time Frame: 1.5 hours
Population: Analyses were conducted for all groups who received a digital assessment combined. Only scores for the first assessment were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Total Sample: IntelliSpace Cognition (ISC): Philips ISC is a Class-II Medical Device in the US and provides objective data regarding cognition via scoring algorithms that HCPs can use to inform diagnostic decision making and treatment planning. It enables tracking cognition over time and offers the possibility of new outcome measures. ISC can be used in a variety of healthcare environments such as neurology and neuropsychology practices.
Arm/Group | Total Sample
Number analyzed (Participants) | 300
units on a scale
  Rey Auditory Verbal Learning Test (score range 0-45, higher score indicates better outcome) | 41.3 (9.5)
  Clock Test Drawing (on scale from 0-22, higher score indicates better outcome) | 17.9 (3.9)
  Clock Test Copy (on scale from 0-22, higher score indicates better outcome) | 19.3 (2.3)
  Rey Osterrieth Complex Figure Test Copy (scale 0-36, higher score indicating better outcome) | 29.1 (6.6)
  Rey Osterrieth Complex Figure Test Recall (scale 0-36, higher score indicating better outcome) | 9.5 (6.3)
  Digit Span forward (number of items correct, range 0-12, higher score indicating better outcome) | 7.8 (2.2)
  Digit Span backward (number of items correct, range 0-12, higher score indicating better outcome) | 6.5 (2.5)
Statistical Analysis 1: Comparison: Total Sample; Test type: Equivalence — Validity and test-retest reliability were explored; p > .05, t-test, 2 sided; Mean Difference (Final Values) = .05; Validity and test-retest reliability were explored

2. Primary Outcome: Scores Digital (ISC) Tests
Description: as for outcome 1
Time Frame: 1.5 hours
Description (as registered): Scores retrieved from all cognitive tests on the ISC platform The cognitive tests included on the ISC platform are commonly used in neuropsychological assessments and measure aspects of executive functioning (TMT A, TMT B, Star Cancellation Test, RAVLT, Letter Fluency Test, Category Fluency Test, ROCFT, Digit Span Forward, Digit Span Backward), processing speed (Star Cancellation Test), working memory (TMT A, TMT B, Star Cancellation Test, Letter Fluency Test, Digit Span Forward, Digit Span Backward), memory (RAVLT), verbal processing (Letter Fluency Test, Category Fluency Test), and visual-spatial processing (RAVLT, ROCFT).
  Star Cancellation Test (completion time divided by number of correct cancellations, higher=worse)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Total Sample
Number analyzed (Participants) | 300
seconds
  Trail Making Test A (in seconds) | 40.9 (12.4)
  Trail Making Test B (in seconds) | 104.7 (55)

3. Primary Outcome: Scores Digital (ISC) Tests
Description: Scores retrieved from all cognitive tests on the ISC platform The cognitive tests included on the ISC platform are commonly used in neuropsychological assessments and measure aspects of executive functioning (TMT A, TMT B, Star Cancellation Test, RAVLT, Letter Fluency Test, Category Fluency Test, ROCFT, Digit Span Forward, Digit Span Backward), processing speed (Star Cancellation Test), working memory (TMT A, TMT B, Star Cancellation Test, Letter Fluency Test, Digit Span Forward, Digit Span Backward), memory (RAVLT), verbal processing (Letter Fluency Test, Category Fluency Test), and visual-spatial processing (RAVLT, ROCFT).
  Star Cancellation Test (completion time divided by number of correct cancellations, higher=worse)
Time Frame: 1.5 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: completion time/number correct words
Arm/Group | Total Sample
Number analyzed (Participants) | 300
completion time/number correct words | .9 (.2)

4. Primary Outcome: Scores Digital (ISC) Tests
Description: as for outcome 1
Time Frame: 1.5 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of words
Arm/Group | Total Sample
Number analyzed (Participants) | 300
number of words
  Letter Fluency Test (sum of correct words in 3 trials, higher score indicating better outcome) | 38.7 (11)
  Category Fluency Test (sum of correct words in 3 trials, higher score indicating better outcome) | 45.9 (9.5)

5. Primary Outcome: Scores From Paper Tests
Description: Scores from paper tests The paper cognitive tests included are the same as the tests included on the ISC platform are commonly used in neuropsychological assessments and measure aspects of executive functioning (TMT A, TMT B, Star Cancellation Test, RAVLT, Letter Fluency Test, Category Fluency Test, ROCFT, Digit Span Forward, Digit Span Backward), processing speed (Star Cancellation Test), working memory (TMT A, TMT B, Star Cancellation Test, Letter Fluency Test, Digit Span Forward, Digit Span Backward), memory (RAVLT), verbal processing (Letter Fluency Test, Category Fluency Test), and visual-spatial processing (RAVLT, ROCFT).
Time Frame: 1.5 hours
Population: Descriptives
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Paper-pencil Group: All groups combined that have received the paper-pencil cognitive tests. Only visit 1 performance is reported.
Arm/Group | Paper-pencil Group
Number analyzed (Participants) | 150
units on a scale
  Rey Auditory Verbal Learning Test (range 0-45, higher score indicating better outcome) | 41.3 (8.1)
  Clock Test Drawing (range 0-12, higher score indicating better outcome) | 8.1 (2.4)
  Clock Test Copy (range 0-12, higher score indicating better outcome) | 9.6 (.7)
  Rey Osterrieth Complex Figure Test Copy (range 0-36, higher score indicating better outcome) | 27.2 (6.8)
  Rey Osterrieth Complex Figure Test Recall (range 0-36, higher score indicating better outcome) | 11.2 (6.1)
  Digit Span forward (number of correct items, range 0-12, higher indicating better outcome) | 8 (2.1)
  Digit Span backward (number of correct items, range 0-12, higher indicating better outcome) | 6.2 (2)

6. Primary Outcome: Scores From Paper Tests
Description: as for outcome 5
Time Frame: 1.5 hours
Description (as registered): Scores from paper tests The paper cognitive tests included are the same as the tests included on the ISC platform are commonly used in neuropsychological assessments and measure aspects of executive functioning (TMT A, TMT B, Star Cancellation Test, RAVLT, Letter Fluency Test, Category Fluency Test, ROCFT, Digit Span Forward, Digit Span Backward), processing speed (Star Cancellation Test), working memory (TMT A, TMT B, Star Cancellation Test, Letter Fluency Test, Digit Span Forward, Digit Span Backward), memory (RAVLT), verbal processing (Letter Fluency Test, Category Fluency Test), and visual-spatial processing (RAVLT, ROCFT).
  Star Cancellation Test (completion time divided by number of correct cancellations, higher=worse)
Population: Descriptives
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Paper-pencil Group
Number analyzed (Participants) | 150
seconds
  Trail Making Test A (in seconds, higher indicating worse outcome) | 33.9 (10.7)
  Trail Making Test B (in seconds, higher indicating worse outcome) | 85 (48.6)

7. Primary Outcome: Scores From Paper Tests
Description: Scores from paper tests The paper cognitive tests included are the same as the tests included on the ISC platform are commonly used in neuropsychological assessments and measure aspects of executive functioning (TMT A, TMT B, Star Cancellation Test, RAVLT, Letter Fluency Test, Category Fluency Test, ROCFT, Digit Span Forward, Digit Span Backward), processing speed (Star Cancellation Test), working memory (TMT A, TMT B, Star Cancellation Test, Letter Fluency Test, Digit Span Forward, Digit Span Backward), memory (RAVLT), verbal processing (Letter Fluency Test, Category Fluency Test), and visual-spatial processing (RAVLT, ROCFT).
  Star Cancellation Test (completion time divided by number of correct cancellations, higher=worse)
Time Frame: 1.5 hours
Population: Descriptives
Measure: Mean (Standard Deviation); unit: completion time/number correct words
Arm/Group | Paper-pencil Group
Number analyzed (Participants) | 150
completion time/number correct words | .8 (.3)

8. Primary Outcome: Scores From Paper Tests
Description: as for outcome 5
Time Frame: 1.5 hours
Population: Descriptives
Measure: Mean (Standard Deviation); unit: number of words
Arm/Group | Paper-pencil Group
Number analyzed (Participants) | 150
number of words
  Letter Fluency Test (sum of correct words during 3 trials, higher indicating better outcome) | 41 (11.9)
  Category Fluency Test (sum of correct words in 3 trials, higher score indicating better outcome) | 46 (9.2)

ADVERSE EVENTS:
Time Frame: For each participant, an assessment took approximately 1.5 hours. Any adverse events during this time period were recorded and reported within 24 hours.
Description: There were no serious adverse events.
Groups:
- Digital / Paper: Participants in this arm first received the digital tests and then the paper tests.
- Paper / Digital: Participants in this arm first received the paper tests and then the digital tests.
- Digital / Digital: Participants in this arm received the digital tests during both assessments.
- Paper / Paper: Participants in this arm received the paper tests during both assessments.
- Digital: Participants in this arm received only one (digital) assessment.
Arm/Group | Digital / Paper | Paper / Digital | Digital / Digital | Paper / Paper | Digital
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/101 | 0/53 | 0/49 | 0/148
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/101 | 0/53 | 0/49 | 0/148
Other Adverse Events (participants affected / at risk) | 0/99 | 0/101 | 0/53 | 0/49 | 0/148

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03801382/Prot_SAP_002.pdf